CLINICAL TRIAL: NCT03175419
Title: BReLLS: A Prospective Belgian Registry on Laparoscopic Liver Surgery
Acronym: BReLLS
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, AHHK, Prof. Dr. Roberto Troisi, University Hospital, Ghent
Other Study IDs: B670201627155
Record Dates: First submitted 2017-05-23; First posted 2017-06-05 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Laparoscopic Liver Surgery
Keywords: laparoscopic liver resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Setting up a Prospective Belgian National Registry of patients undergoing minimally invasive liver resections will allow the constitution of a national network able to get updated information on indication and results. Data will be of great importance for additional scientific projects aimed to clarify the role of minimally invasive approach in surgical liver pathology, especially malignancies.

DETAILED DESCRIPTION:
During recent years we saw over the world a consistent growth of laparoscopic liver surgery (LLS), essentially due to progress of the surgical techniques, technology and diagnostic imaging. During the Louisville conference on LLS (2008) the technique was thoroughly described and defined. One of the most important statements was the promotion of national registries, taking into account the logistics and feasibility problems of randomized trials in this setting. The main purpose to hold a Belgian national registry is to define the role of LLS in our country, looking for short and long-term outcomes, especially in case of liver tumors.

In Belgium approximately 1000 liver resections are performed each year, however, the rate and results of LLS are unknown. The prospective data collection will highlight the role and incidence of LLS. Eventually, the registry will serve as support for scientific projects on different topics.

The evolution of the national practice will be measured by looking to the ratio between laparoscopic and open procedures registered in the electronic CRF (eCRF) in a single center during a time period.

The registration of additional parameters (as per below) will be necessary for comparing outcomes between conventional and laparoscopic techniques.

The registered cases will be recorded prospectively and consecutively.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hepatic resection with minimally invasive approach (laparoscopic and robotic assisted)
* minimum age of > or = 18 years
* Signed informed consent.
* Cysts deroofing
* Laparoscopic resections combined to ablation procedures
* Ablation procedures (RFA, MWA, other)

Exclusion criteria:

* Laparoscopic staging procedures of the liver with/without intraoperative ultrasonography and/or biopsy.
* Solely others therapeutic procedure of the liver (RFA, MWA, PV ligation, etc.)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be observed from the time of recruitment and throughout the hospital stay and will be collected information on vital status until discharge and planned follow-up.
  There is a minimum of 1-year follow-up required. Upon the evolution of patients inclusion and the available resources, we will consider to extend the FU time especially for oncological issues.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Clavien-dindo grade I | 24 month
  Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions.Allowed therapeutic regimens are: drugs as antiemetics, antipyretics, analgetics, diuretics and electrolytes and physiotherapy. This grade also includes wound infections opened at the bedside.
Clavien-dindo grade II | 24 month
  Requiring pharmacological treatment with drugs other than such allowed for grade I complications.
  Blood transfusions and total parenteral nutrition are also included.
Clavien-dindo grade III A and B | 24 month
  Requiring surgical, endoscopic or radiological intervention, intervention not (A) under general anesthesia; intervention under general anesthesia (B)
Clavien-dindo grade IV | 24 month
  Life-threatening complication (including CNS complications)‡ requiring IC/ICU-management
Clavien-dindo grade V | 24 month
  Death of a patient

SECONDARY OUTCOMES:
Mortality | 24 month
  Incidence
Evolution of the laparoscopic approach | 24 month
  Comparison between open and lap procedures in the same center
Assessment of tumor margins | 24 month
  Comparison between R0 and R1 margins
Outcome in HCC and CRLM | 24 month
  Overall and disease free survival calculation for the specific above mentioned pathologies

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Tomassini F, Scuderi V, Berardi G, Dili A, D'Hondt M, Sergeant G, Hubert C, Huysentruyt F, Berrevoet F, Lucidi V, Troisi RI. The practice of laparoscopic liver surgery in Belgium: a national survey. Acta Chir Belg. 2017 Feb;117(1):15-20. doi: 10.1080/00015458.2016.1202478. Epub 2016 Aug 19. PMID 27541973